CLINICAL TRIAL: NCT05235698
Title: Study of Vascular Endothelial Glycocalyx and Ophthalmic Injury in a Single-center, Cross-sectional, Prospective Cohort of Patients With Prolonged Post-COVID-19 Symptoms
Brief Title: Study of Vascular Endothelial Glycocalyx and Ophthalmic Injury, Prospective Cohort of Patients With Prolonged Post-COVID-19 Symptoms
Acronym: GLYCOVLONG
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MMF_2021_24
Record Dates: First submitted 2022-02-10; First posted 2022-02-11 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: COVID-19; Long COVID
Keywords: GlycoCheck; Glycocalix; Ophthalmological effects of long COVID
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with long COVID diagnosis: Ophthalmological examinations performed as part of the care Addition of GlycoCheck for the study
  Interventions: Procedure: Ophthalmological examinations; Procedure: GlycoCheck

INTERVENTIONS:
Procedure: Ophthalmological examinations — Visual acuity, slit lamp examination, eye pressure, retinophotography, indocyanine green retinal angiography, OCT-A( Optical Coherence Tomography- Angiography), adaptive optics, automated visual field
Procedure: GlycoCheck — Evaluation of the glycocalyx of sublingual capillaries with the GlycoCheck :
  A sidestream dark field camera, coupled with GlycoCheck™ software is used to visualize the patient's sublingual microvascularization

SUMMARY:
The glycocalyx is a membrane coat composed of glycoproteins attached to the surface of cell membranes. Recent publications have drawn attention to the potential role of a degradation of the endothelial glycocalyx (a kind of gel that lines all the vessels of the body) during the SARS-CoV-2 (Severe Acute Respiratory Syndrome - coronavirus 2) epidemic.

The work of Yamaoka-Tojo et al. reveals vascular endothelial dysfunction in patients at high risk for developing a severe form of COVID 19. This observation prompts further investigation of vascular endothelial function in SARS-CoV-2-infected patients, and particularly those with long COVID.

As of the end of the first COVID-19 epidemic wave in May 2020, persistence of symptoms several weeks or months after the first manifestations of COVID-19 was described in more than 20% of patients after 5 weeks and in more than 10% after 3 months). The term "long COVID" describes this phenomenon of prolonged symptoms following COVID-19.

The French National Authority for Health has established criteria to identify people with prolonged symptoms after an initial episode of clinically and/or biologically documented COVID-19: an initial symptomatic episode, the presence of at least one of the initial symptoms beyond 4 weeks after the onset of the acute phase of the disease, and initial and prolonged symptoms not explained by another diagnosis not known to be related to COVID-19.

Among the observations reported in patients with long COVID, ophthalmic involvement is poorly described.

A team of ophthalmologists of the Rothschild Foundation has demonstrated (using indocyanine green angiography, adaptive optics and optical coherence tomography techniques) disorders of the choroidal circulation, with abnormalities of the vascular walls, presence of "pachyvessels" and "caverns", in COVID-positive patients hospitalized at 6 months of their hospitalization.

DETAILED DESCRIPTION:
The aim of this study is to extend the exploration of the microvascular system by a microscopic imaging technique of sublingual blood capillaries. The GlycoCheck is a medical device with CE marking. It is the only all-in-one automated system that includes patented software technology embedded in a dedicated computer, a digital video microscope camera, and the calculation of a MicroVascular Health Score™. The video microscope camera is placed under the tongue, showing the live movement of red blood cells as they move through the microvessels. Higher scores indicate a healthier microvascular system. When the transparent glycocalyx lining of the microvascular system is healthy, so are the blood vessels, which are essential for health and vitality. A clinical video microscope detects erythrocytes in the small sublingual blood vessels. Then the GlycoCheck software records, detects and analyzes blood vessels from 5 to 25 µm in diameter. The automatic analysis consists of the detection of the central lumen of each blood vessel and the detection of the outer limits of the erythrocytes. The distance between the red cell column and this outer boundary is identified as the Perfused Boundary Region (PBR). The PBR value is calculated over 3000 individual positions, which makes the measurement results sensitive, but highly reproducible. A higher PBR value corresponds to a proportional decrease in the thickness of the glycocalyx layer. There are 3000 vascular segments per test. These segments process 3,000,000 capillary markers that track the movement of red blood cells and how they interact with the endothelial glycocalyx. Results are provided within minutes of test completion and a microvascular health report is created. This medical device has already been used in numerous clinical studies.

The main objective is to search for associations between possible ocular abnormalities and possible glycocalyx abnormalities evaluated by the GlycoCheck

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of long COVID, namely:

  1. Initial symptomatic episode of COVID-19: Either confirmed by at least one of the following criteria: Positive SARS-Cov-2 PCR (polymerase chain reaction, positive SARS-CoV-2 antigenic test, prolonged anosmia/ageusia of abrupt onset, typical chest CT (computerized tomography) scan (bilateral ground glass pneumonia...), or probable by the association of at least 3 criteria, of sudden onset, in an epidemic context, among: fever, headache, fatigue, myalgia, dyspnea, cough, chest pain, diarrhea, odynophagia. A positive SARS-CoV-2 serology may help in this diagnosis.
  2. Presence of at least one of the initial symptoms beyond 4 weeks after the onset of the acute phase of the disease
  3. Initial and prolonged symptoms not explained by another diagnosis with no known relationship to COVID-19
* Referred for ophthalmologic evaluation to the Rothschild Foundation Hospital
* Expressed consent to participate in the study

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Known allergy to indocyanine green

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with COVID long referred to the Rothschild Hospital for an ophthalmological assessment
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Capillary density (mm/mm²) | Baseline
  Assessed by the GlycoCheck
PBR : Perfused Boundary Region (µm) | Baseline
  Assessed by the GlycoCheck
Capillary velocity of red blood cells (µm/s) | Baseline
  Assessed by the GlycoCheck
Micro Vascular Health Score | Baseline
  Assessed by the GlycoCheck:
  Score from 0 to 10. 10 is the best score for Micro Vascular Health and 0 the worse.
Presence of vascular hyperpermeability | Baseline
  Determined by an ophthalmologist with the images of indocyanine green angiography
Presence of vascular wall abnormalities | Baseline
  Determined by an ophthalmologist with the results of adaptive optics
Presence of vessel dilatation | Baseline
  Determined by an ophthalmologist with the images of OCT (Optical Coherence Tomography)

CONTACTS AND LOCATIONS:
Overall Officials: Martine MAUGET-FAYSSE, MD, Principal Investigator — Rothschild Hospital Foundation
Locations (1):
- Hospital-Foundation Adolphe de Rothschild, Paris, France